CLINICAL TRIAL: NCT05357144
Title: AmbassADDOrs for Health: Supporting Young Women's Health Through Girl-friendly Drug Vendors
Brief Title: AmbassADDOrs for Health Study
Acronym: ADDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); Health for a Prosperous Nation (Other); RTI International (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH124516 (NIH); R01MH124516 (NIH)
Record Dates: First submitted 2022-04-18; First posted 2022-05-02 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections
Keywords: HIV self-testing; Human-centred design; Adolescent health; Contraception; Drug shops
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial; Catchment areas will be randomly assigned 1:1 to intervention or comparison arms (n=60-70 intervention drug shops; ~3-4 drug shops per area) using a constrained approach to ensure balance in key covariates.
Who Masked: Investigator
Masking Description: No blinding or masking to treatment status throughout the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug shops, also known as Accredited Drug Dispensing Outlets (ADDOs), owners or staff (Experimental): All drug shopkeepers in intervention areas (within Shinyanga or Mwanza) will be invited to participate in Malkia Klabu, a loyalty card program. Consenting drug shops in intervention areas should be willing and able to keep records of referrals and sexual and reproductive health (SRH) product distribution given to AGYW through the use of Maisha Meds during the one month run-in period.
  Interventions: Behavioral: Loyalty card program at drug shops & supply of HIVST and SRH products
- Shopkeepers in control arm for comparison area (Placebo Comparator): Drug shopkeepers, staff and/or owners as part of the control arm will receive standard HIV training, guidance on referring AGYW to proximal HIV care, and HIVST for free distribution to AGYW.
  Interventions: Behavioral: Comparison drug shops

INTERVENTIONS:
Behavioral: Loyalty card program at drug shops & supply of HIVST and SRH products — Consenting drug shops will receive:
  * training on Malkia Klabu implementation;
  * HIVST training (same as comparison drug shops);
  * procedures for referring to youth-friendly HIV/SRH services;
  * a monthly supply of HIVST reserved for free distribution to AGYW, with "free" price stickers and pre-packaged with referral information; and
  * reimbursement for SRH products given to AGYW (e.g., birth control pills).
  Arms: Drug shops, also known as Accredited Drug Dispensing Outlets (ADDOs), owners or staff
Behavioral: Comparison drug shops — Consenting drug shops in the comparison arm catchment areas will have access to the Maisha Meds inventory management application system for offline digital recording of HIVST, HIVST kits earmarked for free to AGYW, guidance on HIV care referral plan to facilitate linkage to nearby health facilities for AGYW. These control drug shops will not participate in Malkia Klabu (Queen Club) program implementation.
  Arms: Shopkeepers in control arm for comparison area

SUMMARY:
The goal of the study is to evaluate Malkia Klabu ("Queen Club") in Tanzania, a loyalty program intervention that creates adolescent girls and young women (AGYW)-friendly drug shops where AGYW can access HIV prevention services and contraception.

DETAILED DESCRIPTION:
The investigators will conduct a cluster-randomized controlled trial of the Malkia Klabu intervention in 40 health facility catchment areas (n=60-70 intervention drug shops; ~3-4 drug shops per area) in the Shinyanga and Mwanza regions of Tanzania, plus a mixed-methods, implementation science study to pinpoint supply-side factors influencing effectiveness (e.g., implementation models, intervention fidelity, shop characteristics).

Malkia Klabu is a loyalty card program derived from a youth participatory process with human centered design. Young women earn punches on the Malkia Klabu loyalty card when they make drug shop purchases that upon accrual can be used towards prizes of increasing value. When joining, young women receive a free HIV self test kit (HIVST) as an opt out sign-up gift, are invited to interact with a physical display of sexual and reproductive health products, including HIVST, and may elect to view videos on a tablet computer about the program, HIVST, and contraception. The back of the card displays discreet symbols representing sensitive products available at the shop (e.g., HIVST, oral contraception). Club members can ask for or point to the product that they want on the card and receive it for free in a discreet bag. Referrals are provided to youth-friendly services at a nearby catchment area health facility for HIV testing, treatment and care, and/or contraception.

ELIGIBILITY:
The primary unit of analysis are the wards, and within them, the drug shops who will be enrolled based on the following inclusion criteria:

Inclusion Criteria:

* Wards with no greater than 3 public health facilities;
* Wards with no less than 4 drug shops;
* Wards with health facilities that were greater than 20 KM from a primary or secondary road; and
* Drug shop owners and staff in Shinyanga and Mwanza Regions of Tanzania who are aged 18 or older;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative HIV diagnoses among 15-24 year old females | 12-15 months
  Cumulative HIV-positive tests among 15-24 year old females at 12-15 months from routinely collected health facility data, disaggregated by sex and age, aggregated to the catchment area level.
Antenatal care registrations by 15-24 year old females | 12-15 months
  Cumulative antenatal care registrations among 15-24 year old females at 12-15 months from routinely collected health facility data, disaggregated by age, aggregated to the catchment area level.

SECONDARY OUTCOMES:
ART initiation among newly diagnosed AGYW | 12-15 months
  Data on ART initiation abstracted from routinely collected health facility data, disaggregated by sex and age, aggregated to the catchment area level.
Distribution of HIVST to AGYW | 12-15 months
  Distribution of HIVST to AGYW will be documented in Maisha Meds, a point of sales inventory system to be used by participating drug shops in both arms. This will be a continuous variable with a lower limit of zero and an undefined upper limit and is the simple count of all HIVSTs distributed to AGYW who visit the shops.
Distribution contraception to AGYW | 12-15 months
  Distribution of contraception to AGYW will be documented in Maisha Meds, a point of sales inventory system to be used by participating drug shops in both arms. This will be a continuous variable with a lower limit of zero and an undefined upper limit and is the simple count of the combined total number of oral contraceptive pills, emergency contraception, and condoms sold to AGYW who visit the shops.
Program exposure | 12-15 months
  Self-reported data from AGYW on exposure to Malkia Klabu (if any) will be collected during an endline survey. This will be a proportion defined as the number of AGYW who report ever receiving a Malkia Klabu card (i.e. enrolling) as the numerator over the total number of AGYW interviewed. The values will range from 0-100%.
Recent HIV testing | 12-15 months
  Self-reported data from AGYW on recent HIV testing (if any) will be collected during an endline survey. This will be a proportion defined as the number of AGYW who report testing for HIV in the last 6 months as the numerator over the total number of AGYW interviewed. The values will range from 0-100%.
Recent pregnancy testing | 12-15 months
  Self-reported data from AGYW on recent pregnancy testing (if any) will be collected during an endline survey. This will be a proportion defined as the number of AGYW who report taking a pregnancy test in the last 6 months as the numerator over the total number of AGYW interviewed. The values will range from 0-100%.
Unmet need for contraception | 12-15 months
  Self-reported data from AGYW on contraceptive preferences, desires, and use (if any) will be collected during an endline survey. Unmet need is defined as the number of women who do not want to get pregnant but are not using a method of birth control and are sexually active. We will use the collected data to create a variable where the numerator is the number of women not using a method of birth control and do not desire to get pregnant over the total number of sexually active women.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny X Liu, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- Tanzania (2):
  - Mwanza Province, Mwanza
  - Shinyanga Province, Shinyanga

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make the data and associated documentation available to users upon request and only under a data-sharing agreement with the study team that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The SP, SAP, and ICF will be made available on the Open Science Framework (OSF) within 12 months recruitment.
  Study results will be posted to OSF and Clinical Trials within 12 months of completion of data collection.
Access Criteria: Everything posted to OSF and Clinical Trials will be made publicly available.

REFERENCES:
- [Background] Hunter LA, McCoy SI, Rao A, Mnyippembe A, Hassan K, Njau P, Mfaume R, Liu JX. Designing drug shops for young women in Tanzania: applying human-centred design to facilitate access to HIV self-testing and contraception. Health Policy Plan. 2021 Nov 11;36(10):1562-1573. doi: 10.1093/heapol/czab084. PMID 34313728
- [Background] Liu J, Prach LM, Treleaven E, Hansen M, Anyanti J, Jagha T, Seaman V, Ajumobi O, Isiguzo C. The role of drug vendors in improving basic health-care services in Nigeria. Bull World Health Organ. 2016 Apr 1;94(4):267-75. doi: 10.2471/BLT.15.154666. Epub 2016 Feb 3. PMID 27034520
- [Background] Peters DH, Mirchandani GG, Hansen PM. Strategies for engaging the private sector in sexual and reproductive health: how effective are they? Health Policy Plan. 2004 Oct;19 Suppl 1:i5-i21. doi: 10.1093/heapol/czh041. PMID 15452011
- [Background] Corroon M, Kebede E, Spektor G, Speizer I. Key Role of Drug Shops and Pharmacies for Family Planning in Urban Nigeria and Kenya. Glob Health Sci Pract. 2016 Dec 28;4(4):594-609. doi: 10.9745/GHSP-D-16-00197. Print 2016 Dec 23. PMID 28031299
- [Background] Rutta E, Liana J, Embrey M, Johnson K, Kimatta S, Valimba R, Lieber R, Shekalaghe E, Sillo H. Accrediting retail drug shops to strengthen Tanzania's public health system: an ADDO case study. J Pharm Policy Pract. 2015 Sep 25;8:23. doi: 10.1186/s40545-015-0044-4. eCollection 2015. PMID 26413304
- [Background] Sieverding M, Schatzkin E, Shen J, Liu J. Bias in Contraceptive Provision to Young Women Among Private Health Care Providers in South West Nigeria. Int Perspect Sex Reprod Health. 2018 Mar 1;44(1):19-29. doi: 10.1363/44e5418. PMID 30028307
- [Derived] Mnyippembe A, Sheira LA, McCoy SI, Njau PF, Packel LJ, Hassan K, Solorzano-Barrera C, Maokola W, Kang Dufour MS, Sabasaba A, Liu J. Supporting young women's health through girl-friendly drug vendors in Lake Zone, Tanzania: protocol for the AmbassADDOrs for Health cluster-randomised controlled trial. BMJ Open. 2024 Jun 8;14(6):e078755. doi: 10.1136/bmjopen-2023-078755. PMID 38851225